CLINICAL TRIAL: NCT04566367
Title: Detection Rate by Blue Laser Imaging (BLI) of Secondary or Early Squamous Head and Neck Cancer in Patients Undergoing Elective Percutaneous Endoscopic Gastrostomy (PEG)
Brief Title: Blue Laser Imaging (BLI) for Detection of Secondary Head and Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Georg Dultz (Other)
Responsible Party: Sponsor-Investigator, Georg Dultz, Record Keeper, Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: JWGUHMED1-011
Record Dates: First submitted 2018-12-02; First posted 2020-09-28 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-06

CONDITIONS: Head Neck Cancer; Esophageal Cancer; Gastrostomy
Keywords: esophageal cancer; Blue laser imaging; percutaneous endoscopic gastrostomy; head neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a prospective randomised mono centric study with a one to one allocation in two different treatment arms.
Who Masked: Participant
Masking Description: The participants don't know which arm they were allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard White Light Imaging (Active Comparator): In this group the participants will be examined by white light endoscopy first and secondly with blue laser imaging technique during the same gastroscopy.
  Interventions: Diagnostic Test: blue laser imaging
- Blue Light Imaging (Experimental): In this group the participants will be examined by blue laser imaging technique first and secondly with standard white light during the same gastroscopy.
  Interventions: Diagnostic Test: blue laser imaging

INTERVENTIONS:
Diagnostic Test: blue laser imaging — The intervention is the push on demand activation of blue laser imaging technique during gastroscopy.

SUMMARY:
This study wants to focus on Carcinoma detection rates with blue laser imaging (BLI) for participants with head-neck cancer who need a percutaneous endoscopic gastrostomy (PEG). BLI is a new imaging technique that can easily be used within a standard gastroscopy.

DETAILED DESCRIPTION:
Head-Neck cancers are a significant burden all around the world. Patients suffering from one tumor are at high risk for a second cancer or another precancerous lesion. Before or during cancer treatment a PEG is needed to maintain a sufficient calories intake. PEG is established by performing a standard gastroscopy.

This randomised study wants to compare the detection rates of standard white light endoscopy compared to the additional use of blue laser imaging for second cancers or precancerous lesions in participants presenting for PEG establishment.

ELIGIBILITY:
Inclusion Criteria:

* All participants with the need of PEG due to head neck cancers or esophageal carcinoma

Exclusion Criteria:

* Minors, pregnant women, contraindication for endoscopy, contraindications for establishment of a PEG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Detection rate of a second cancer or precancerous lesions | The time frame is during the PEG insertion (approximately 15min)
  The detection rates for malignant or premalignant lesions in participants with head neck tumors will be compared when using BLI and white light endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Mireen Friedrich-Rust, Professor, Principal Investigator — Goethe University
Locations (1):
- Klinikum der J. W. Goethe-Universität, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No